CLINICAL TRIAL: NCT05724498
Title: A Randomized Clinical Trial Comparing Brief and Standard Cognitive-Behavioral Therapies for Insomnia in Veterans
Brief Title: Brief Versus Standard Cognitive Behavioral Therapy for Insomnia in Veterans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Finger Lakes Healthcare System (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3840-R; 1I01RX003840-01A2 (NIH)
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Insomnia
Keywords: Insomnia; Cognitive-Behavioral Therapy for Insomnia; Functional Health; Mental Health; Veterans
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Veterans randomized to either brief (4 session) or full (6 session) Cognitive-Behavioral Therapy for Insomnia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive-Behavioral Therapy for Insomnia (CBT-I) (Active Comparator): Compare two behavioral interventions for insomnia
  Interventions: Behavioral: Brief CBT-I; Behavioral: Standard CBT-I
- Standard Cognitive-Behavioral Therapy for Insomnia (CBT-I) (Active Comparator): Standard VA 6 session version of CBT-I
  Interventions: Behavioral: Brief CBT-I; Behavioral: Standard CBT-I

INTERVENTIONS:
Behavioral: Brief CBT-I — 4 session CBT-I
Behavioral: Standard CBT-I — Standard VA 6 session CBT-I

SUMMARY:
Insomnia is a common condition in Veterans, with prevalence rates as high as 53% among treatment-seeking Veterans. Chronic untreated insomnia is associated with increased risk for functional impairment, psychiatric illness, suicidal ideation, unhealthy lifestyles, and decreased quality of life. Cognitive-Behavioral Therapy for Insomnia (CBT-I) is recognized as the first-line treatment for insomnia. Despite its proven efficacy, CBT-I is not always readily provided and/or accessible to Veterans. To address these limitations, behavioral sleep medicine specialists have endeavored to streamline CBT-I through development of time-shortened variations of CBT-I. Although these modifications show promise for advancing care and access, studies comparing brief treatments to standard CBT-I have yet to be performed. This investigation will therefore compare a 4-session brief CBT-I to VA standard 6-session CBT-I to evaluate whether a brief intervention can provide comparable benefits to sleep, functional, and psychiatric outcomes in Veterans with insomnia.

DETAILED DESCRIPTION:
Veterans seen in VA primary care and mental health clinics commonly present with complaints of sleep disturbance, especially insomnia. For example, in a cross-sectional study examining sleep disorders among Veterans seeking care through the Veterans Health Administration between 2000-2010, sleep apnea (47%) and insomnia (26%) were the most commonly diagnosed conditions. In a study of 375 Operation Enduring Freedom/Operation Iraqi Freedom Veterans, 45% reported extended time spent trying to fall asleep (> 30 minutes), 21% reported reduced total sleep times (< 4.5 hours), and 56% reported being awake in bed more than 15% of the night. Similarly, in another observational study of 5,552 Veterans, 57.2% of the sample population was found to have insomnia disorder. This sample also was at high-risk for a host of clinical disorders, including PTSD, TBI, and pain; all of which showed higher rates of insomnia.

Cognitive Behavioral Therapy for Insomnia (CBT-I) is a multi-component intervention that features sleep restriction, stimulus control, sleep hygiene education, cognitive therapy, and can include relaxation techniques. CBT-I is recognized as the first-line treatment for chronic insomnia and is effective in Veterans, however, limitations to use still remain. In recent years advances in treatment approaches have attempted to streamline CBT-I by focusing on delivery of specific treatment components, reducing number of treatment sessions, and/or use of technologies that provide for ease of dissemination and implementation. Brief Cognitive-Behavioral Therapy for Insomnia (bCBT-I) represents one such empirically tested brief intervention which may decrease patient burden through reduced sessions needed to achieve treatment goals and through use of hybrid treatment administration (i.e., in-person and telemedicine).

To better inform both clinical practice and future research, this investigation proposes to assess the comparative effectiveness of bCBT-I to VA standard CBT-, with several overarching goals: 1) in a randomized clinical trial (RCT), evaluate the equivalence (non-inferiority) of bCBT-I to VA standard CBT-I; 2) evaluate the impact of these treatment approaches on functional rehabilitation outcomes; 3) evaluate the impact of these treatment approaches on psychiatric symptomatology; and 4) in an exploratory fashion, determine which patient factors best predict success or failure with a given treatment as a means of developing insomnia phenotypes that might be used diagnostically to match patient characteristics and type of treatment to help optimize clinical outcomes (i.e., a "personalized medicine" approach to treatment).

The investigation timeline consists of four parts: 1) baseline assessment of sleep, functional, and psychiatric outcome measures; 2) randomization and assignment to either CBT-I or bCBT-I; 3) post-treatment assessment; and 4) 3-month follow-up assessment. Over 40 months of recruitment this study will enroll and randomize 180 Veterans on a 1:1 ratio (CBT-I:bCBT-I= 90:90) from VA primary care and mental health clinics at two Centers of Excellence sites (VA San Diego Healthcare System and Finger Lakes VAMC Healthcare System). For the primary study aim, one-sided mean difference testing will be conducted with the noninferiority margin added to the null value. Secondary analyses will utilize structural equation modeling to evaluate how CBT-I and bCBT-I influence functional and psychosocial outcomes. The Exploratory aim will utilize moderation analyses to better understand for whom either CBT-I and/or bCBT-I might be more effective.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of insomnia as classified by the (a) Diagnostic and Statistical Manual of Mental Disorders-5 (DSM 5) which includes daytime impairment in functioning for > 3 months and occurring at least 3 nights per week and (b) subjective sleep disturbance defined by an Insomnia Severity Index (ISI) score >7 at intake
2. Meets current DSM 5 criteria for a comorbid mental health disorder
3. No formal therapist guided treatment with brief or standard Cognitive-Behavioral Therapy for Insomnia within the past 2 years
4. on stable medication regimen for at least 4 weeks prior to enrollment in study.

Exclusion Criteria:

1. History of a acute or unstable neurological disorder(s), dementia, or premorbid IQ <70
2. Schizophrenia, psychotic disorder, and/or bipolar disorder
3. Suicidality more than "medium risk" as determined by the VA Comprehensive Suicide Risk Assessment
4. Sleep disturbances other than insomnia (e.g., untreated obstructive sleep apnea, periodic limb movements, narcolepsy, and/or circadian-based sleep disruptions)
5. alcohol and/or substance use disorder for 90 days prior to intake, but past history of alcohol and/or substance use is not exclusionary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) scores from pretreatment to follow-up | Week 0 (baseline) and Week 20 (follow-up)
  Measure of insomnia severity (0-24; higher score equals worse insomnia)

SECONDARY OUTCOMES:
Change in Functional Outcomes of Sleep Questionnaire 10 (FOSQ-10) | Week 0 (baseline) and Week 20 (follow-up)
  Self-report measure of the impact of sleep on daytime functioning (five domains scored 1-4; lower score equals more impairment)
Change in Pittsburgh Sleep Quality Index (PSQI) scores from pretreatment to follow-up | Week 0 (baseline) and Week 20 (follow-up)
  Self-report measure of general sleep disturbance (0-21 scale; higher score equals greater sleep disturbance)
Change in WHO Disability Assessment Schedule (WHODAS 2.0) | Week 0 (baseline) and Week 20 (follow-up)
  Self-report measure of disability and functioning (six domains scored 1-5; summary score from 0-100 with higher score equals greater disability)
Change in Brief Inventory of Psychosocial Functioning (B-IPF) | Week 0 (baseline) and Week 20 (follow-up)
  Self-report measure of PTSD related functional impairment (0-6 scale; items summed so that higher score equals greater impairment)
Change in PTSD Checklist for DSM 5 (PCL-5) | Week 0 (baseline) and Week 20 (follow-up)
  Self-report measure of symptoms in relation to a traumatic event (score 0-80; scores greater than 33 equal clinically significant level of symptoms)
Change in Patient Health Questionnaire 9 (PHQ 9) | Week 0 (baseline) and Week 20 (follow-up)
  Self-report measure of depressive symptoms (0-27 scale; higher scores equal more depressive symptoms)
Change in Generalized Anxiety Disorder Scale 7 (GAD-7) | Week 0 (baseline) and Week 20 (follow-up)
  Self-report measure of anxiety symptoms (0-21 scale; higher scores equal more anxiety symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Henry J. Orff, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (2):
- United States (2):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Finger Lakes Healthcare System, Canandaigua, NY, Canandaigua, New York

IPD SHARING:
Plan to Share IPD: No